CLINICAL TRIAL: NCT06061042
Title: The Effect of Timed-Restricted Eating on Insulin Sensitivity, De Novo Lipogenesis and Liver Fat in Subjects With Obesity and Insulin Resistance
Brief Title: Effect of Timed-Restricted Eating on Metabolic Health
Acronym: TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Diabetesfonds (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Mireille JM Serlie, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL79197.018.21
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Non-Alcoholic Fatty Liver Disease; Insulin Resistance
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early time-restricted eating (Experimental): * 50% of daily calories at breakfast, 35% at lunch and 15% at dinner. 85% of calories consumed in 6h, i.e., between 7AM and 1PM.
  * Eating period, 10h (7AM-5PM); fasting period, 14h; Breakfast between 7 and 8 AM; lunch between 12 AM and 1 PM; dinner between 4 and 5 PM.
  Interventions: Behavioral: Early time restricted eating
- Late time-restricted eating (Experimental): * 15% of daily calories at breakfast, 35% at lunch and 50% at dinner. 85% of calories consumed in 6h, i.e., between 2PM and 8PM.
  * Eating period, 10h (10AM-8PM), fasting period, 14h; Breakfast between 10 and 11 AM; lunch between 2 and 3 PM; dinner between 7 and 8 PM.
  Interventions: Behavioral: Late time restricted eating

INTERVENTIONS:
Behavioral: Early time restricted eating — Subjects will follow an isocaloric diet, designed by a dietician. The eating window for the early-TRE group is between 7 AM - 5 PM
  Other Names: early-TRE
  Arms: Early time-restricted eating
Behavioral: Late time restricted eating — Subjects will follow an isocaloric diet, designed by a dietician. The eating window for the late-TRE group is between 10 AM - 8 PM
  Other Names: late-TRE
  Arms: Late time-restricted eating

SUMMARY:
We aim to determine the effect of combined isocaloric time restricted eating and meal timing on metabolic health, liver fat, functional brain networks, inflammation, and sleep pattern/quality in subjects with obesity and insulin resistance.

DETAILED DESCRIPTION:
Obesity is an alarming global health issue, with increasing prevalence. Obesity leads to a vast array of disorders, including dyslipidemia, the accumulation of intrahepatic triglycerides (IHTG), multiorgan insulin resistance and type 2 diabetes mellitus. In addition, disruption of the circadian rhythm (circadian misalignment), which is associated with irregular eating schedules, is an important risk factor for the development of obesity, IHTG and type 2 diabetes mellitus. Time restricted eating (TRE) is a form of intermittent fasting, in which the daily eating period is restricted. The beneficial effect of this type of diet might relate to adequate synchronization of food intake and fasting to the internal rhythm of the circadian tissue clocks, improving metabolic handling of nutrients and metabolic flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent;
* BMI > 30kg/m^2;
* Insulin resistance, as defined by fasting plasma insulin > 62 pmol/L and/or prediabetes, as defined by fasting plasma glucose > 5.3 and < 7.0 mmol/L;
* Stable weight for 3 months prior to study inclusion
* For women, 1 year after last menstrual cycle

Exclusion Criteria:

* Use of any medication, except for those related to treatment of metabolic syndrome;
* Any medical condition interfering with study outcomes or design;
* History of any psychiatric disorder, including eating disorders;
* Performing shift work
* Performing intensive sports (>3 hours/week);
* Smoking;
* Drugs abuse or alcohol abuse (>3 units/day);
* Contraindication for MRI;
* Known lactose/gluten intolerance;
* Known soy, egg, milk or peanut allergy;
* Childhood onset of obesity

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will use the Oral Minimal Model Method in conjunction with a Mixed Meal Tolerance Test (MMTT) to quantitatively evaluate insulin sensitivity. Concentrations of insulin, glucose, and C-peptide will be measured during the course of the MMTT to serve as the requisite inputs for the model. The output is in dl/kg/min/uU/ml.

SECONDARY OUTCOMES:
Change in plasma insulin | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Fasted and stimulated insulin (pmol/L) will be measured during MMTT
Change in plasma glucose | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Fasted and stimulated glucose (mmol/L) will be measured during MMTT
Change in intrahepatic fat | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  To quantify the intrahepatic fat content, a single voxel 1H-MRS (magnetic resonance spectroscopy) will be used. Relative fat content will be expressed as the ratio of the fat peak over the cumulative fat and water peak. This will also be corrected for T2 relaxation.
Change in beta cell function (C-peptide) | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Fasted and stimulated C-peptide (nmol/L) will be measured during MMTT
Change in insulin aignaling | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Biopsies will be taken from skeletal muscle and subcutaneous fat to measure key proteins in the insulin signalling pathway (Western blots)
Change in glucose variability | Baseline 1 to week 4 for intervention 1, Baseline 2 to week 12 for intervention 2
  In our study, we will deploy Continuous Glucose Monitors (CGMs) to acquire an in-depth understanding of glucose variability in participants throughout the course of the intervention. These monitors gauge glucose concentrations in the interstitial fluid (mmol/L), serving as a reliable proxy for blood glucose levels. This approach will enable us to assess key metrics such as mean, minimum and maximum glucose levels.
De novo lipogenesis | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Fasted and stimulated de novo lipogenesis (DNL) will be measured during the MMT as 2H incorporation into fatty acids following deuterated water (2H2O) administration
Immunological markers | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will conduct immune cell phenotyping on whole blood samples to identify and categorize various immune cell types. Additionally, we will assess immune cell function and metabolism in isolated peripheral blood mononuclear cells (PBMCs). Inflammatory markers will also be assessed in serum samples to provide a comprehensive overview of immune and inflammatory status.
Physical activity | Baseline 1 to week 4 for intervention 1, Baseline 2 to week 12 for intervention 2
  Physical activity will be assessed via accelerometry. Accelerometry represents the magnitude of acceleration in any direction, over a predefined epoch.
Functional brain activity | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  Brain activation maps and functional connectivity will be assessed by blood oxygen dependent signals in the resting state and after visual food cues using functional magnetic resonance imaging (fMRI).
Psychological factor - Food Craving | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will use the General Food Cravings Questionnaire (G-FCQ) to evaluate the frequency and intensity of food cravings among participants. The scoring for the G-FCQ ranges between 21 and 105, with higher scores indicative of more pronounced food craving tendencies.
Psychological factor - Eating behaviour | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will utilize the Dutch Eating Behavior Questionnaire (NVE) to assess and categorize the eating behaviors and tendencies of our participants. The NVE discerns three distinct eating styles: emotional eating, external eating, and restrained eating. A higher score within a specific style suggests a predominant inclination towards that particular eating behavior.
Psychological factor - Hunger scale | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will employ a nine-question visual analogue scale (VAS) to assess hunger. Each question will be scored 0-100.
Psychological factor - Food addiction | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will use the Yale Food Addiction Scale 2.0 (YFAS 2.0) to assess addictive behaviours. The YFAS 2.0 is designed in accordance with the DSM-5 criteria, and its scoring system mirrors the number of DSM-5 criteria fulfilled indicative of addiction.
Psychological factor - Impulsiveness | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will use the Barratt Impulsiveness Scale (BIS) to scale impulsiveness towards food. This will help us understand how impulsivity might influence dietary behaviour. The score ranges from 30-120 and a higher score leans towards greater impulsivity.
Psychological factor - Chronotype | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  To determine natural sleep-wake patterns, we will use the Munich Chronotype Questionnaire (MCTQ). This tool offers a comprehensive understanding of sleep behaviors, revealing a chronotype.
Subject experience with intervention | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We will employ a semi-structured oral interview as part of our qualitative approach to understand our participants' experience and adherence to the intervention.
Delay discounting computational task | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  The delay discounting task aids in understanding the decision-making processes that might contribute to overeating and poor food choices. In this task, we will be able to measure the ability of each individual to delay immediate gratification for a greater future reward.
Iowa gambling computational task | Baseline 1 and week 4 for intervention 1; Baseline 2 and week 12 for intervention 2
  We use the Iowa gambling task to assess decision-making and risk-reward sensitivity. Participants choose cards from four decks, each with different reward and punishment rates, aiming to maximize their winnings. We use this task to study risk taking and impulsive behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille JM Serlie, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No